CLINICAL TRIAL: NCT06079541
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of JMKX003142 Tablets Administered Randomly, Double-blind, Placebo-controlled Single and Multiple Times in Healthy Adult Subjects, as Well as the Effects of Randomized, Open, and Two Cycle Crossover Foods
Brief Title: Phase 1 Clinical Study of JMKX003142 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jemincare (Industry)
Collaborators: Zhejiang Hangyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: JY-JM-035-101
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-07

CONDITIONS: Safety and Tolerability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- JMKX003142 SAD experimental group (Experimental): Participants will be randomized into 7 cohorts to receive single oral dose of JMKX003142 on Day 1. The doses in each cohort will be escalated based on the safety and pharmacokinetics (PK) / Pharmacodynamics (PD) data of the previous cohort.
  Interventions: Drug: JMKX003142 will be administered orally
- JMKX003142 MAD experimental group (Experimental): Participants will be randomized into 3 cohorts to receive orally once -daily of JMKX003142 for 7 consecutive days. The second cohort will be escalated based on the safety and pharmacokinetics (PK)/ Pharmacodynamics (PD) data of the previous cohort.
  Interventions: Drug: JMKX003142 will be administered orally
- JMKX003142 FE experimental group (Experimental): Participants will receive 2 Sequence regimens, with a washout period between treatments.
  Interventions: Drug: JMKX003142 will be administered orally
- Placebo in Cohorts 1 to 7 (Experimental): Participants in Cohorts 1 to 7 will receive single oral dose of matching placebo on Day 1.
  Interventions: Drug: Placebo in Cohorts 1 to 7
- Placebo in 3 Cohorts (Experimental): Participants in 3 Cohorts will receive orally once -daily of matching placebo for 7 consecutive days.
  Interventions: Drug: Placebo in 3 Cohorts

INTERVENTIONS:
Drug: JMKX003142 will be administered orally — oral once
  Other Names: JMKX003142
  Arms: JMKX003142 SAD experimental group
Drug: JMKX003142 will be administered orally — oral once
  Other Names: JMKX003142
  Arms: JMKX003142 MAD experimental group
Drug: JMKX003142 will be administered orally — oral once
  Other Names: JMKX003142
  Arms: JMKX003142 FE experimental group
Drug: Placebo in Cohorts 1 to 7 — oral once
  Other Names: Matching placebo will be administered orally
  Arms: Placebo in Cohorts 1 to 7
Drug: Placebo in 3 Cohorts — oral once
  Other Names: Matching placebo will be administered orally
  Arms: Placebo in 3 Cohorts

SUMMARY:
Phase I clinical study to evaluate the safety, tolerability, and pharmacokinetic characteristics of JMKX003142 tablets administered randomly, double-blind, placebo-controlled single and multiple times in healthy adult subjects, as well as the effects of randomized, open, and two cycle crossover foods

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-45 years (including boundary values)
2. Able to sign a written informed consent form
3. Physical examination, clinical laboratory examination value, Virology examination, vital signs and 12 lead ECG examination are confirmed by the researcher to be normal or abnormal without clinical significance
4. The subjects have a thorough understanding of the study content, process, and potential adverse effects, and are willing to complete the study according to the requirements of the experimental protocol

Exclusion Criteria:

1. Had or currently have serious clinical diseases related to circulatory system, respiratory system, digestive system, nervous system, endocrine system, blood lymphatic system, genitourinary system or psychiatry, as well as habitual constipation, gastrointestinal bleeding history, which is judged to be inappropriate for the study by the investigators
2. Participants in any other clinical study within 3 months prior to the first administration of this study
3. The investigators believe that the subject has other factors that are not suitable for participating in this experiment
4. Pregnant or lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of the Adverse Events that are related to the single dose treatment | from baseline to Day 18
  single dose safety
Number of the Adverse Events that are related to the multiple dose treatment from | from baseline to Day 24
  multiple dose safety

CONTACTS AND LOCATIONS:
Overall Officials: Xuening li, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China